CLINICAL TRIAL: NCT03999086
Title: Thromboelastography-guided Fluid Management in Spinal Surgery: A Prospective Analysis
Brief Title: Thromboelastography-Guided Fluid Management in Spinal Surgery
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jamal McClendon, Jr., Principal Investigator, Mayo Clinic
Other Study IDs: 17-006702
Record Dates: First submitted 2018-05-07; First posted 2019-06-26 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Spinal Fusion
MeSH Terms: interventions — Methods; Thrombelastography; Control Groups; Point-of-Care Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Traditional evaluation/standard-of-care evaluation of patients undergoing multi-level spinal fusion surgery. These patients will receive point-of-care laboratory testing.
  Interventions: Other: Control Group
- Intervention arm: Utilization of TEG for decision-making regarding intra-operative transfusion in major spinal reconstruction surgery.
  Interventions: Procedure: Intervention

INTERVENTIONS:
Procedure: Intervention — We will utilize thromboelastography to discern when to transfuse blood products in the setting of multi-level spinal fusion
  Other Names: Thromboelastography
  Groups: Intervention arm
Other: Control Group — Laboratory analysis to guide transfusion
  Other Names: Point of care testing
  Groups: Control Group

SUMMARY:
The Researchers are trying to evaluate whether using a blood test called thromboelastogram (TEG) to manage patients undergoing multi-level spinal fusion surgery will reduce complications after surgery compared with the standard practices.

DETAILED DESCRIPTION:
Multi-level instrumented spinal fusions represent an important treatment modality for degenerative scoliosis and sagittal malalignment. These surgeries remain a significant physiologic burden with high blood loss and long operative times. Thromboelastography provides a quantitative measure for blood product transfusion surrounding procedures. We aim to utilize thromboelastography to guide transfusions for multi-level spinal instrumentation. This two-arm, randomized, non-blinded prospective analysis will clarify reduced transfusion requirements for TEG-arm compared to non-TEG arm. We will also evaluate postoperative outcomes at the 1 year time-point.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing elective multi-level spinal fusion for sagittal malalignment, multi-level spondylolisthesis, multi-level lumbar spinal stenosis, and adult degenerative scoliosis with ages between 18-89

Exclusion Criteria:

* patients with tumors, infection, or trauma

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Mayo Clinic receiving a multi-level spinal fusion surgery.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Estimated Blood Loss | post operative approximately 1 day
  Amount of blood loss measured in units of cc(mL)
Volume of transfused packed red blood cells | post operative approximately 1 day
  Amount of transfused packed red blood cells measured in units of cc(mL)
Adverse Events | One year
  Number of adverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Jamal McClendon, Jr., MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials